CLINICAL TRIAL: NCT06499701
Title: Volume Kinetics of Fluid Resuscitation With 30 ml/kg Ringer Lactate in Early Sepsis
Brief Title: Volume Kinetics of Fluid Resuscitation in Early Sepsis
Status: Recruiting | Type: Observational
Sponsor: Institutul de Urgenţă pentru Boli Cardiovasculare Prof.Dr. C.C. Iliescu (Other)
Responsible Party: Principal Investigator, Balan Ion Cosmin, Principal Investigator, Institutul de Urgenţă pentru Boli Cardiovasculare Prof.Dr. C.C. Iliescu
Other Study IDs: 17736
Record Dates: First submitted 2024-07-07; First posted 2024-07-12 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Fluid and Electrolyte Imbalance
Keywords: volume kinetics; sepsis; volume resuscitation; crystalloid; Ringer's Lactate
MeSH Terms: conditions — Sepsis | interventions — Ringer's Lactate; Crystalloid Solutions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Ringer's Lactate: Adult patients admitted in the intensive care unit (ICU) with sepsis, as defined by the Sepsis-3 criteria and exhibiting sepsis-induced hypoperfusion prior to the administration of adequate volume resuscitation (i.e., 30 ml/kg crystalloid).
  Interventions: Drug: Ringer's Lactate

INTERVENTIONS:
Drug: Ringer's Lactate — Ringer's Lactate is administered at a dose of 30ml/kg, with the first 20ml/kg given at a constant rate over the initial 30 minutes, followed by a 30-minute pause, and then an additional 10ml/kg over the next 15 minutes, completing the infusion within 75 minutes.
  Other Names: Crystalloid

SUMMARY:
The recommended volume resuscitation for patients with early sepsis-induced hypoperfusion is at least 30 ml/kg of crystalloid administered within the first three hours. However, this standardized approach does not account for individual patient variability and lacks personalization. Additionally, the effects of administering 30 ml/kg on intercompartmental fluid shifts between the plasma and interstitial compartments remain unclear. This study aims to describe the volume kinetics of administering 30 ml/kg of Ringer's Lactate in patients with early sepsis-induced hypoperfusion within the first three hours.

DETAILED DESCRIPTION:
Adult patients admitted to the intensive care unit (ICU) with sepsis, as defined by the Sepsis-3 criteria, and exhibiting sepsis-induced hypoperfusion prior to receiving adequate volume resuscitation (i.e., 30 ml/kg of crystalloid), are administered Ringer's Lactate at a dose of 30 ml/kg. The initial 20 ml/kg is infused at a constant rate over the first 30 minutes, followed by a 30-minute pause, with an additional 10 ml/kg administered over the subsequent 15 minutes, completing the infusion within 75 minutes.

Up to 180 minutes post-infusion, no other fluids (e.g., gelatin, albumin) are administered except for antibiotics, sedatives, or vasoactive substances as needed. Ideally, only one catecholamine (e.g., norepinephrine) is administered. The volume and quantity of these substances are recorded. Arterial blood samples are collected for blood gas analysis, including hemoglobin levels. Urinary output is measured at 30, 60, and 180 minutes, and any blood loss, other than the 1.5 ml per sample collected, is quantified during hemoglobin monitoring. Additionally, urinary creatinine concentration is determined from urine samples collected at baseline.

The hemodilution data are utilized as input into a three-compartment model with microconstants for fluid redistribution and excretion.

ELIGIBILITY:
Inclusion Criteria:

A diagnosis of sepsis, as defined by the Sepsis-3 criteria and exhibiting sepsis-induced hypoperfusion prior to the administration of adequate volume resuscitation:

* hypotension requiring norepinephrine to maintain a mean arterial blood pressure (MAP) either predefined by the clinician or at 65 mm Hg or higher and/or
* a serum lactate level >2 mmol/L (18mg/dL) and/or
* acute oliguria defined as urine output <0.5mL/kg/hr and/or
* mottled skin and/or
* capillary refill time > 3 seconds.

Exclusion Criteria:

* Administration of at least 1 L of IV fluid in the last 6 hours prior to screening. All crystalloids, colloids and blood products that the patient has received are counted.
* Known pregnancy.
* Competing causes of lactic acidosis including: seizures within 3 hours of enrollment, use of linezolid or metformin or anti-retrovirals at the time of enrollment, carbon monoxide or cyanide poisoning, highly suspected or known ischemic bowel, and known mitochondrial disorders.
* End-stage renal disease that requires chronic dialysis.
* Concurrent haemorrhagic or obstructive shock.
* Increased risk of fluid intolerance:

  * Echocardiographic evidence of moderate or severe left ventricular systolic dysfunction.
  * Echocardiographic evidence of moderate or severe right ventricular systolic dysfunction.
  * Hypoxemia index < 200 mmHg or sonographic evidence of bilateral B or C profile.
  * Abdominal compartment syndrome.
* Post-cardiac arrest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted in the intensive care unit (ICU) with sepsis, as defined by the Sepsis-3 criteria and exhibiting sepsis-induced hypoperfusion prior to the administration of adequate volume resuscitation.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Plasma Volume | 180 minutes after the start of the Ringer's Lactate infusion
  Plasma volume (ml) was determined using a three-compartment kinetic model with five rate constants (k12, k21, k23, k32 and k10) and a scaling factor (Vc, central volume) that relates dilution to volume. This model was applied to the dependent variables, which included frequently measured plasma dilution and urinary excretion.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hahn, Professor, Study Chair — Karolinska Institutet: Stockholm, SE (Department of Clinical Sciences, Danderyd Hospital) Employment; Serban-Ion Bubenek-Turconi, Professor, Study Director — "Prof CC Iliescu" Emergency Institue for Cardiovascular Diseases
Locations (2):
- Romania (2):
  - Fundeni Clinical Institute, Bucharest, București
  - "Prof CC Iliescu" Emergency Institue for Cardiovascular Diseases, Bucharest